CLINICAL TRIAL: NCT05966259
Title: Management of Childhood Obesity in the Context of Primary Health Care: an Intensive Multi-level Intervention
Brief Title: Management of Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adaliene Versiani M. Ferreira (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundacion MAPFRE (Other)
Responsible Party: Sponsor-Investigator, Adaliene Versiani M. Ferreira, Doctor, Federal University of Minas Gerais
Organization: Federal University of Minas Gerais (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 39508720.6.0000.5149
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Childhood Obesity; Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Intervention Group: intensive multilevel intervention, with a minimum of 26 contact hours, for a period of 5 months. The children will be re-evaluated in the eighth month (three months after intervention) and in the eleventh month (six months after intervention). The monthly activities were composed of four weekly contacts: Individual Attendance, Food and Nutrition Education (at home), Group Food and Nutrition Education in the basic health unit and Telephone monitoring. There will be five monthly themes: food, physical activity, sedentary behavior, sleep, and mental health. The children in the Control Group were followed in a similar way, observing the activities so that they did not exceed 26 hours of contact, during the 5 months.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group- Intensive Multilevel Intervention (Other): Intervention Group: intensive multilevel intervention, with a minimum of 26 contact hours, for a period of 5 months. The children will be re-evaluated in the eighth month (three months after intervention) and in the eleventh month (six months after intervention). The monthly activities were composed of four weekly contacts: Individual Attendance, Food and Nutrition Education (at home), Group Food and Nutrition Education in the basic health unit and Telephone monitoring. There will be five monthly themes: food, physical activity, sedentary behavior, sleep, and mental health.
  Interventions: Other: Intervention Group- Intensive Multilevel Intervention
- Control Group (Other): The children in the Control Group were followed in a similar way, observing the activities so that they did not exceed 26 hours of contact, during the 5 months.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Intervention Group- Intensive Multilevel Intervention — intensive multilevel intervention, with a minimum of 26 contact hours, for a period of 5 months. The children will be re-evaluated in the eighth month (three months after intervention) and in the eleventh month (six months after intervention). The monthly activities were composed of four weekly contacts: Individual Attendance, Food and Nutrition Education (at home), Group Food and Nutrition Education in the basic health unit and Telephone monitoring. There will be five monthly themes: food, physical activity, sedentary behavior, sleep, and mental health.
  Other Names: Intensive Multilevel Intervention
  Arms: Intervention Group- Intensive Multilevel Intervention
Other: Control Group — The children in the Control Group were followed in a similar way, observing the activities so that they did not exceed 26 hours of contact, during the 5 months.
  Arms: Control Group

SUMMARY:
The significant increase in the prevalence of obesity can also be attributed to various social changes, in which the environment (political, economic, social, cultural), and not only the individual and his choices, takes a strategic place in the analysis of the problem and proposed interventions. The food environment can influence the choice and consumption of foods that promote obesity, such as ultra-processed foods (UPA). It is suggested that to intervene to effectively change behavior and eating habits, intensive interventions are needed that consider multiple levels that include the family, school, and community rather than one-off interventions that may not be effective in changing behavior and lifestyle. Regarding the family environment, parents or guardians can assist in the adoption of obesity-related behavioral patterns. It is known that the context of Primary Health Care (PHC) is ideal for actions to prevent diseases and promote children's health, since the PHC professional team is closest to the reality of life of the child, family, and community. We emphasize the importance of this study from the perspective of treatment of childhood obesity, in order to generate scientific evidence and practical subsidies for the implementation of interventions focused not only on the individual, but also in the context of the Unified Health System (SUS). The hypothesis of the study is that there will be a decrease in the consumption of ultra-processed foods (UPA) among children, aged 6 to 10 years, living with obesity and who are treated in primary health care. In addition to encouraging healthy habits such as physical activity and the consumption of in natura and minimally processed foods. The management of childhood obesity is one of the priority topics on the national agenda of SUS's food, nutrition, and health promotion policies.

ELIGIBILITY:
Inclusion Criteria:

* child classified as obesity by values equal to or greater than z-score +2 for BMI/age

Exclusion Criteria:

* children with severe mental disorders
* children on weight loss medication and with comorbidities associated with obesity
* children participating in any diet and physical activity program for weight loss/maintenance
* parents/guardians who do not agree to participate and do not sign the informed consent form

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Consumption of ultra-processed foods | After 5 months
  10% reduction in consumption of ultra-processed foods

SECONDARY OUTCOMES:
BMI Z score by age | After completion of the study (12 months)
  Reduce and/or maintain BMI Z score by age

CONTACTS AND LOCATIONS:
Overall Officials: Larissa L Mendes, Doctor, Principal Investigator — UFMG
Locations (1):
- Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil